CLINICAL TRIAL: NCT02637817
Title: MRI-based Biomarkers for the Prognosis Judgement of Punctate White Matter Lesions in Neonates: a Longitudinal Multicenter Study
Brief Title: MRI-based Biomarkers for Predicting Punctate White Matter Lesions in Neonates
Acronym: PWML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); General Hospital of Ningxia Medical University (Other); Xijing Hospital (Other); Shengjing Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zunyi Medical College (Other); Shaanxi Provincial People's Hospital (Other); Baoji Central Hospital (Other); Children's Hospital of Fudan University (Other); Hainan People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016YFC0100300
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Brain Diseases; Amblyopia; Brain Damage, Chronic; Cerebral Palsy
MeSH Terms: conditions — Brain Diseases; Amblyopia; Brain Damage, Chronic; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control Group: Neonates with no evidence of brain lesions on conventional MRI.
- Patients Group: Neonates with PWML diagnosed by conventional MRI.

SUMMARY:
As a common white matter (WM) disease in preterm neonates, punctate white matter lesion (PWML) frequently leads to the abnormalities of brain development (e.g. the motor, visual and auditory disorders), even to cerebral palsy (CP) and amblyopia during childhood. However, it is lack of certain methods in identifying the prognosis of PWML. Through using various advanced MRI techniques, neuro-behavioral and visual assessments, a multicenter longitudinal study would be conducted to follow-up the PWML neonates with varying spatial-position and degree lesions. Through tracking the variations in WM microstructures from neonate period to childhood (2 years old and 3 years old), this study aims to explore (1) the potential relations between varying PWMLs and motor and visual disorders (2) the relations between WM MRI-metrics and neurodevelopmental assessment results, and thus determine the early biomarkers to identify CP and amblyopia.

ELIGIBILITY:
Inclusion Criteria:

-(1) Age: 1-28 days (2) PWML (3) High quality MRI scan

Exclusion Criteria:

-(1) Congenital malformations, infections, metabolic disorders, intraventricular hemorrhage (2) Neonates of mothers with gestational diabetes, hypertension, hypoglycemia and history of alcohol

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PWML and non-PWML neonates
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral Palsy | At age 2
  The enrolled subjects who will be diagnosed as cerebral palsy by clinical examination at age 2.

SECONDARY OUTCOMES:
Amblyopia or movement disorder | At age 3
  The enrolled subjects who will be diagnosed as amblyopia or movement disorder by clinical examination at age 3.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wang M, Liu H, Liu C, Li X, Jin C, Sun Q, Liu Z, Zheng J, Yang J. Prediction of adverse motor outcome for neonates with punctate white matter lesions by MRI images using radiomics strategy: protocol for a prospective cohort multicentre study. BMJ Open. 2019 Apr 3;9(4):e023157. doi: 10.1136/bmjopen-2018-023157. PMID 30948562